CLINICAL TRIAL: NCT02495402
Title: Substance Abuse Treatment to HIV Care (SAT2HIV): The Motivational Interviewing-based Brief Intervention (MIBI) Experiment
Brief Title: Substance Abuse Treatment to HIV Care (SAT2HIV): The Motivational Interviewing-based Brief Intervention Experiment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SAT2HIV; R01DA038146 (NIH)
Record Dates: First submitted 2015-07-06; First posted 2015-07-13 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Substance Use
MeSH Terms: conditions — Substance-Related Disorders | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention: Control (No Intervention): No Intervention
- Motivational Interviewing (Experimental): A brief interview intervention for substance abuse
  Interventions: Behavioral: Motivational Interviewing

INTERVENTIONS:
Behavioral: Motivational Interviewing — Participants assigned to the experimental condition receive a single 20-30 minute motivational interviewing-based brief intervention for substance use.
  Arms: Motivational Interviewing

SUMMARY:
To test the effectiveness of a single 20-30 minute motivational interviewing-based brief intervention for substance use within HIV/AIDS settings.

DETAILED DESCRIPTION:
The Substance Abuse Treatment to HIV care (SAT2HIV) project, a Type 2 Effectiveness-Implementation Hybrid Trial, seeks to address this gap in services by providing new knowledge regarding the effectiveness of brief intervention (BI) for substance use within community-based HIV/AIDS service settings, as well as new knowledge regarding how to address the well-documented underutilization of evidence-based practices in real-world settings. The specific aims of this project are: Aim 1: To experimentally test the effectiveness of a motivational interviewing-based BI for substance use within community-based HIV/AIDS service organizations, relative to usual care (UC). Aim 2: To experimentally test the effectiveness of adding an organizational-level implementation intervention called Implementation & Sustainment Facilitation (ISF) to enhance the effectiveness of the implementation strategy currently used by SAMHSA-funded Addiction Technology Treatment Centers (ATTCs; i.e., online introductory training, 2-day training workshop, ongoing feedback and coaching).

ELIGIBILITY:
Inclusion Criteria:

* Have HIV/AIDS.
* Be 18 years of age or older.
* Acknowledges use of at least one substance within the past 28 days and endorse 2+ substance use disorder symptoms during the past 12-months.
* Provide signed and dated assurance of consent.

Exclusion Criteria:

* Are unable to speak English.
* Are unwilling to allow brief intervention sessions to be audio recorded.
* Are unwilling to participate in the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 827 (Actual)
Dates: Start 2015-07-08 (Actual); Primary Completion 2017-12-28 (Actual); Study Completion 2018-03-25 (Actual)

PRIMARY OUTCOMES:
Days of Primary Substance Use | 4 weeks post randomization
  Days of Primary Substance Use - A continuous measure (ranges from 0 - 28) that is based on a question that asks participants to report how many days during the past 28 days they used their primary substance.
Number of Substance-related problems | 4 weeks post randomization
  Number of Substance-related problems - A continuous measure (ranges from 0 - 11) that represents the sum of the number of 11 DSM-V substance use disorder symptoms participants report having occured during the past 28 days.
Times engaging in risky behaviors | 4 weeks post randomization
  Times engaging in risky behaviors - A continuous measure (no specified range) that is based on a question that asks participants to report how many times during the past 28 days they engaged in unprotected sex, IV drug use, or needle sharing.
Days of Substance Use Treatment | 4 weeks post randomization
  Days of Substance Use Treatment - A continuous measure (no specified range) that represents the sum of the number of days participants report going to residential treatment, outpatient treatment, or self-help group meetings during the past 28 days.
ART Medication Adherence | 4 weeks post randomization
  ART Medication Adherence - A continuous measure (ranges from 0 -28) that is based on a question that asks participants to report how many days during the past 28 days that they have missed at least one dose of their HIV medications.

SECONDARY OUTCOMES:
Urgency to Change | 4 weeks post randomization
  Urgency to Change - A continuous measure (ranges from 0 - 20) that represents the sum of two questions that ask participants to use a Likert-type scale where 0 equals "Not at all" and 10 equals "The highest level possible" to indicate their urgency during the past 4 weeks to a) reduce their use of their primary substance and b) completely stop using their primary substance.
Intentions to Change | 4 weeks post randomization
  Intentions to Change - A continuous measure (ranges from 0 - 20) that represents the sum of two questions that ask participants to use a Likert-type scale where 0 equals "Not at all" and 10 equals "The highest level possible" to indicate their intentions during the past 4 weeks to a) reduce their use of their primary substance and b) completely stop using their primary substance.
Commitment to Change | 4 weeks post randomization
  Commitment to Change - A continuous measure (ranges from 0 - 20) that represents the sum of two questions that ask participants to use a Likert-type scale where 0 equals "Not at all" and 10 equals "The highest level possible" to indicate their commitment during the past 4 weeks to a) reduce their use of their primary substance and b) completely stop using their primary substance.
Self-Efficacy to Change | 4 weeks post randomization
  Self Efficacy for Change - A continuous measure (ranges from 0 - 20) that represents the sum of two questions that ask participants to use a Likert-type scale where 0 equals "Not at all" and 10 equals "The highest level possible" to indicate their confidence during the past 4 weeks to a) reduce their use of their primary substance and b) completely stop using their primary substance.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan R Garner, PhD, Principal Investigator — RTI International
Locations (39):
- United States (39):
  - HIV Care Directions, Phoenix, Arizona
  - Foothill AIDS Project, Claremont, California
  - AIDS Services Foundation, Orange County, Irvine, California
  - AIDS Project Los Angeles, Los Angeles, California
  - Shanti, San Francisco, California
  - AIDS Project Greater Danbury, Inc., Danbury, Connecticut
  - AIDS Connecticut, Inc, Hartford, Connecticut
  - Delaware HIV Consortium, Wilmington, Delaware
  - The Women's Collective, Washington D.C., District of Columbia
  - Project Response, Inc., Melbourne, Florida
  - Live Forward (AIDS Athens), Athens, Georgia
  - Champaign-Urbana Public Health District (Collaborating Organization), Champaign, Illinois
  - The Project of the Quad Cities (Collaborating Organization), Davenport, Iowa
  - AIDS Volunteers, Inc. (AVOL), Lexington, Kentucky
  - Southwest Louisiana AIDS Council, Lake Charles, Louisiana
  - AIDS Project Worcester, Worcester, Massachusetts
  - Health Emergency Lifeline Programs (Collaborating Organization), Detroit, Michigan
  - Community Health Awareness Group (Collaborating Organization), Detroit, Michigan
  - Community AIDS Resources and Education Services (Collaborating Organization), Kalamazoo, Michigan
  - Minnesota AIDS Project (Collaborating Organization), Minneapolis, Minnesota
  - Burrell Behavioral Health (Collaborating Organization), Springfield, Missouri
  - Doorways (Collaborating Organization), St Louis, Missouri
  - Places for People (Collaborating Organization), St Louis, Missouri
  - Project ARK, St Louis, Missouri
  - St. Louis Effort for AIDS (Collaborating Organization), St Louis, Missouri
  - Nebraska AIDS Project (Collaborating Organization ), Omaha, Nebraska
  - Southern NH HIV/AIDS Task Force, Nashua, New Hampshire
  - Caracole House (Collaborating Organization), Cincinnati, Ohio
  - ARC Ohio (Collaborating Organization), Columbus, Ohio
  - HIV Alliance, Eugene, Oregon
  - AID Upstate, Greenville, South Carolina
  - Chattanooga CARES, Chattanooga, Tennessee
  - Nashville CARES, Nashville, Tennessee
  - Panhandle AIDS Support Organization, Amarillo, Texas
  - Triangle Area Network, Beaumont, Texas
  - AIDS Foundation Houston, Houston, Texas
  - Alamo Area Resource Center, San Antonio, Texas
  - Utah AIDS Foundation, Salt Lake City, Utah
  - Vermont CARES, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ford JH 2nd, Gilson AM, Maurer MA, Hoffman KA, Garner BR. A peek behind the curtain: exploring coaching styles within the implementation and sustainment facilitation (ISF) strategy in the substance abuse treatment to HIV care study. Implement Sci Commun. 2021 Dec 20;2(1):140. doi: 10.1186/s43058-021-00246-2. PMID 34930497
- [Derived] Garner BR, Gotham HJ, Tueller SJ, Ball EL, Kaiser D, Stilen P, Speck K, Vandersloot D, Rieckmann TR, Chaple M, Martin EG, Martino S. Testing the effectiveness of a motivational interviewing-based brief intervention for substance use as an adjunct to usual care in community-based AIDS service organizations: study protocol for a multisite randomized controlled trial. Addict Sci Clin Pract. 2017 Nov 17;12(1):31. doi: 10.1186/s13722-017-0095-8. PMID 29149914